CLINICAL TRIAL: NCT05770973
Title: The Effect of Eyelid Patching After Anterior Lector Reinsertion and Blepharoplasty on Edema, Hematoma, Scar Formation and Ocular Surface Irritation
Brief Title: Effect of Eyelid Patching After Ptosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augenklinik LMU (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-304
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Ptosis, Eyelid
Keywords: Ptosis, Blepharoplasty, Eyelid surgery
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Intervention Model Description: randomized for compression dressing or none
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression dressing (Active Comparator): Randomized, eyes were patched with a compression dressing after surgery.
  Interventions: Other: Compression dressing (build by Kompressen, gauze swabs, Nobamed Paul Danz AG, Wetter, Germany and NOBALUMENAL® - steril, eye pad, Nobamed Paul Danz AG, Wetter, Germany
- No Compression dressing (No Intervention): Randomized, eyes were not patched with a dressing.

INTERVENTIONS:
Other: Compression dressing (build by Kompressen, gauze swabs, Nobamed Paul Danz AG, Wetter, Germany and NOBALUMENAL® - steril, eye pad, Nobamed Paul Danz AG, Wetter, Germany — Compression dressing after ptosis surgery
  Arms: Compression dressing

SUMMARY:
The goal of this randomized, controlled, observer-blinded study is to compare the effect of compression dressing after ptosis surgery.

The main question it aims to answer are:

Effect of dressing on edema, hematoma, scar formation, ocular surface irritation and postoperative pain.

Patients are randomized after surgery for compression dressing or not. Results are scored by a blinded observer.

type of study: clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Ptosis

Exclusion Criteria:

* kongenital ptosis, pre-surgery, trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
hematoma | First postoperative day until 8 weeks after surgery
  degree of hematoma postoperatively. Ranked by a blinded observer on a four point rating scale (0=none, 1=mild, 2=moderate, 3=severe) using phtographies of the patients eyes.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schuh, Principal Investigator — Augenklinik LMU
Locations (1):
- Augenklink LMU, München, Germany

IPD SHARING:
Plan to Share IPD: No
Date will be shared on request.